CLINICAL TRIAL: NCT04913090
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) of XZP-5610 Tablets Following Single- and Multiple-ascending Doses (SAD/MAD) and Food Effects in Healthy Subjects.
Brief Title: A Phase I Clinical Trial of XZP-5610 Tablets in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5610-1-001
Record Dates: First submitted 2021-05-24; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A-experimental (Experimental): Single Ascending Dose (SAD) phase
  Interventions: Drug: XZP-5610 Tablet (for Part A)
- Part A-placebo (Placebo Comparator): Single Ascending Dose (SAD) phase
  Interventions: Drug: Placebo to match XZP-5610 Tablet (for Part A)
- Part B-experimental (Experimental): multiple ascending dose (MAD) phase
  Interventions: Drug: XZP-5610 Tablet (for Part B)
- Part B-placebo (Placebo Comparator): multiple ascending dose (MAD) phase
  Interventions: Drug: Placebo to match XZP-5610 Tablet (for Part B)
- Part C1-experimental (Experimental): Food Effect (FE) phase
  Interventions: Drug: XZP-5610 Tablet （for "Part C1"）; Drug: XZP-5610 Tablet for "Part C2"
- Part C2-experimental (Experimental): Food Effect (FE) phase
  Interventions: Drug: XZP-5610 Tablet （for "Part C1"）; Drug: XZP-5610 Tablet for "Part C2"

INTERVENTIONS:
Drug: XZP-5610 Tablet (for Part A) — Tablet(s) administered orally once daily for 1 Day
  Other Names: 5610
  Arms: Part A-experimental
Drug: Placebo to match XZP-5610 Tablet (for Part A) — Tablet(s) administered orally once daily for 1 Day
  Other Names: 5610 Placebo
  Arms: Part A-placebo
Drug: XZP-5610 Tablet (for Part B) — Tablet(s) administered orally once daily for 14 Days
  Other Names: 5610
  Arms: Part B-experimental
Drug: Placebo to match XZP-5610 Tablet (for Part B) — Tablet(s) administered orally once daily for 14 Days
  Other Names: 5610 Placebo
  Arms: Part B-placebo
Drug: XZP-5610 Tablet （for "Part C1"） — Tablet(s) administered fasted orally once daily for 1 Day
  Other Names: 5610
  Arms: Part C1-experimental; Part C2-experimental
Drug: XZP-5610 Tablet for "Part C2" — Tablet(s) administered after a high-fat meal orally once daily for 1 Day
  Other Names: 5610
  Arms: Part C1-experimental; Part C2-experimental

SUMMARY:
This study will consist of 3 parts: Part A - Single Ascending Dose (SAD) phase, Part B - multiple ascending dose (MAD) phase, and Part C - Food Effect (FE) phase.

DETAILED DESCRIPTION:
Part A and Part B studies were designed as single-center, randomized, double-blind, placebo-controlled, dose-escalation trials to assess the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profiles of single and multiple oral doses of XZP-5610 tablets in healthy adult subjects, and exploring preliminary food effects (non-high-fat meals) in the Part B study. Part C is a single-center, randomized, open, 2×2 crossover design designed to assess the foodeffects on PK of a single oral dose of XZP-5610 tablets in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males or females aged 18 to 60 years (inclusive).
2. Body weight ≥ 50 kg for males and ≥ 45 kg for females; body mass index (BMI) in the range 19.0-28.0 kg/m2 for the non-obese group and in the range of 28.1 -35.0 kg/ 2 for the obese group (inclusive, BMI=weight/height2).
3. No plans to have children within the last 6 months, no plans to donate sperm/egg, and willing to use effective contraception within 6 months after the end of dosing
4. No clinically significant vital signs, physical examination, laboratory tests, or ECG or chest radiograph findings.
5. Subjects understand and comply with the study procedures, voluntarily participate, and sign an Informed Consent Form.

Exclusion Criteria:

1. History or presence of severe systemic diseases such as endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic epilepsy) abnormalities.
2. History of clinically significant ECG abnormalities or family history of long QT syndrome (grandparents, parents and siblings)

   Part A:

   Any of the following was regarded as a criterion for exclusion:
   1. Confirmation of QTcF ≥ 450 ms by repeated measurements;
   2. Confirmation of QRS duration > 120 ms by repeated measurements;
   3. Confirmation of PR interval > 200 ms by repeated measurements;
   4. Findings that lead to difficulties in QTc measurement or difficult interpretation of QTc data;
   5. History of other risk factors for Torsades de Pointes tachycardia (e.g., heart failure, hypokalemia, family history of long QT syndrome);
   6. Presence of uncorrected hypokalemia or hypomagnesemia.

   Parts B and C:

   Any of the following was regarded as a criterion for exclusion:
   1. Family history of long QT syndrome (grandparents, parents and siblings);
   2. Resting QTcF ≥ 450 ms (males) or ≥ 460 ms (females) during the screening or baseline period.
3. Subjects with a known or suspected history of allergy to the test drug or its adjuvant components, or a history of clinically significant severe allergy (e.g., food, drug, latex allergy), or a history of atopic allergic disease (asthma, urticaria, eczematous dermatitis)
4. History of dysphagia or any gastrointestinal disorder affecting drug absorption at screening, including history of frequent nausea or vomiting of any etiology, history of irregular gastrointestinal motility such as habitual diarrhea, constipation or bowel pre-excitation syndrome, or history of major gastrointestinal surgery (e.g., gastrectomy, gastrointestinal anastomosis, bowel resection, gastric bypass, gastric division, or gastric banding)
5. History of pancreatic injury or pancreatitis at screening, or significantly elevated blood amylase (> 1.5 x ULN)
6. History of urinary tract obstruction or presence of urinary voiding difficulties at screening.
7. History of cancer (malignancy) at the time of screening.
8. Positive test results for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or syphilis antibody
9. History of significant drug abuse within 12 months prior to screening or positive urine drug screening
10. Regular alcohol consumption within 3 months prior to screening, consuming more than 3 alcoholic drinks per day (one drink is approximately equal to: beer 354 mL/12 ounces, wine 118 mL/4 ounces, or distilled spirits 29.5 mL/1 ounce), or evidence of alcohol abuse and excessive consumption as evidenced by alcohol breath test at screening (subjects who consume 4 alcoholic beverages per day may be enrolled at the investigator's (enrollment is at the discretion of the investigator).
11. History of smoking within 3 months prior to screening, or a positive urine nicotine test at screening, or who cannot give up smoking throughout the study period
12. Excessive daily intake of coffee, tea, cola, energy drinks, or other caffeinated beverages within 3 months prior to screening, with excess defined as more than 6 servings (one servingis approximately equal to 120 mg of caffeine).
13. Major surgery, or donation or loss of blood over 400 mL within 3 months prior to administration.
14. Participation in other clinical trials and treatment with investigational productinvestigational product within 3 months prior to administration.
15. Taken any prescription, over-the-counter, nutraceutical, herbal or proprietary Chinese medicine within 4 weeks prior to administration (or less than 5 half-lives of the drug from the start of the trial).
16. Women who are pregnant or breastfeeding, or of childbearing potential who are not using effective non-hormonal contraception (intrauterine device (IUD), barrier method with spermicide, or surgical sterilization, etc.) or are unwilling to continue using these methods during the trial until 6 months after discontinuation; men of childbearing potential who are unwilling to use physical methods of contraception during the trial until 6 months after discontinuation.
17. Systolic blood pressure ≥ 140 mmHg or < 90 mmHg, and/or diastolic blood pressure ≥ 90 mmHg or < 50 mmHg at screening or prior to dosing
18. Heart rate < 50 or > 100 beats/min at screening or prior to dosing.
19. The estimated glomerular filtration rate (eGFR) < 90 ml/min/ 1.73m2 at screening based on the Modification of Diet in Renal Disease Study (MDRD) formula (see Appendix 1 for calculation formula).
20. At screening, the liver function tests of non-obese group showed any measure of aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), or total bilirubin> upper limit of normal (ULN); the liver function tests of obese group showed AST, ALT, or ALP> 1.5 × ULN, or total bilirubin> ULN.
21. Fasting triglycerides > 200 mg/dL (2.27 mmol/L) at screening.
22. Fasting glucose > 5.6 mmol/L in the non-obese group and > 6.1 mmol/L or glycosylated hemoglobin (HbA1c) ≥ 6.5% in the obese group at screening.
23. Those who could not tolerate blood sample collection.
24. Subjects who are deemed by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-03-04 (Estimated); Study Completion 2022-03-04 (Estimated)

PRIMARY OUTCOMES:
Cmax | Single dose：Day1-Day4 , Multi dose: Day1,Day2,Day7,Day10,Day14-Day17，Food Effect:Day1-Day4,Day8-Day11
Tmax | Single dose：Day1-Day4 , Multi dose: Day1,Day2,Day7,Day10,Day14-Day17，Food Effect:Day1-Day4,Day8-Day11
AUClast | Single dose：Day1-Day4 , Multi dose: Day1,Day2,Day7,Day10,Day14-Day17，Food Effect:Day1-Day4,Day8-Day11
AUCinf | Single dose：Day1-Day4 , Multi dose: Day1,Day2,Day7,Day10,Day14-Day17，Food Effect:Day1-Day4,Day8-Day11
T1/2 | Single dose：Day1-Day4 , Multi dose: Day1,Day2,Day7,Day10,Day14-Day17，Food Effect:Day1-Day4,Day8-Day11
CL/F | Single dose：Day1-Day4 , Multi dose: Day1,Day2,Day7,Day10,Day14-Day17，Food Effect:Day1-Day4,Day8-Day11
Vz/F | Single dose：Day1-Day4 , Multi dose: Day1,Day2,Day7,Day10,Day14-Day17，Food Effect:Day1-Day4,Day8-Day11
Subject incidence of adverse events for XZP-5610 versus placebo | From drug administration to study completion. Single dose：15 days , Multi dose: 42 days，Food Effect: 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Dongyang Liu, Doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No